CLINICAL TRIAL: NCT02951208
Title: Transcranial Direct Current Stimulation Coupled With Virtual Rehabilitation for Negative Symptoms in At-Risk Youth
Brief Title: tDCS Coupled With Virtual Rehabilitation for Negative Symptoms in At-Risk Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, George Foussias, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 039-2016
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Clinical High Risk for Psychosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS + Active VR (Experimental): Active tDCS over the left DLPFC (30 minutes) combined with active VR motivation training (60 minutes), administered 3 times per week for 4 weeks.
  Interventions: Device: Active tDCS; Behavioral: Active VR Motivation Training
- Sham tDCS + Sham VR (Sham Comparator): Sham tDCS over the left DLPFC (30 minutes) combined with sham VR motivation training (60 minutes), administered 3 times per week for 4 weeks.
  Interventions: Device: Sham tDCS; Behavioral: Sham VR Motivation Training

INTERVENTIONS:
Device: Active tDCS — Active anodal tDCS over the left DLPFC, administered for 30 minutes, three times per week for four weeks.
  Other Names: Active Transcranial Direct Current Stimulation
  Arms: Active tDCS + Active VR
Behavioral: Active VR Motivation Training — Active computerized treatment with a virtual reality-based motivation training program, administered for 60 minutes, three times per week for four weeks.
  Arms: Active tDCS + Active VR
Device: Sham tDCS — Sham anodal tDCS over the left DLPFC, administered for 30 minutes, three times per week for four weeks.
  Other Names: Sham Transcranial Direct Current Stimulation
  Arms: Sham tDCS + Sham VR
Behavioral: Sham VR Motivation Training — Sham computerized training in a virtual reality-based environment, administered for 60 minutes, three times per week for four weeks.
  Arms: Sham tDCS + Sham VR

SUMMARY:
Negative symptoms, which include the loss of motivation, social withdrawal and reduced emotional expression are prominent in youth at clinical high risk (CHR) for psychosis. These negative symptoms lead to significant functional impairment and enduring disability in these youth. At present, there are no established treatments for negative symptoms. Recent evidence from independent studies, however, suggests two promising novel treatment approaches for negative symptoms, transcranial direct current stimulation (tDCS), and computerized remediation strategies. The primary aim of this study is to evaluate if tDCS combined with a virtual reality-based computerized remediation (VR) is effective for treating negative symptoms in CHR youth, thereby mitigating the enduring functional disability these symptoms cause.

DETAILED DESCRIPTION:
Negative symptoms, which include amotivation, social withdrawal and diminished emotional expression are prominent in youth at clinical high risk (CHR) for psychosis. Negative symptoms lead to significant functional impairment and enduring disability in these youth regardless of subsequent conversion to psychosis. At present, there are no established treatments for negative symptoms. Recent evidence from independent studies, however, suggests two promising novel treatment approaches for negative symptoms, transcranial direct current stimulation (tDCS), and computerized remediation strategies, both of which have revealed significant therapeutic effects on negative symptoms in schizophrenia (SZ). tDCS involves delivery of a low intensity continuous electrical field to the frontal cortex. tDCS is very safe and well tolerated, and is currently being investigated as a treatment for several psychiatric disorders. tDCS is also Health Canada approved for the treatment of major depressive disorder. The primary aim of this randomized controlled trial is to evaluate if tDCS combined with a virtual reality-based computerized remediation (VR), administered three times per week for four weeks, is effective for treating negative symptoms in CHR youth, thereby mitigating the enduring functional disability these symptoms cause.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 16 and 30;
2. meet CHR criteria for a psychosis risk syndrome determined by the Structured Interview for Prodromal Symptoms (SIPS);
3. have a Scale of Prodromal Symptoms (SOPS) negative subscale (SOPS-Neg) score of > 11, with at least one negative symptom of at least moderate severity (i.e., ≥ 3)

Exclusion Criteria:

1. meet criteria for a current or lifetime psychotic disorder;
2. have an IQ < 70;
3. a history of seizures or clinically significant neurological disorder that may contribute to prodromal symptoms.
4. have been involved in another treatment study in the past 4 weeks.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-10; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Scale of Prodromal Symptoms - Negative Subscale (SOPS-Neg) | 8 weeks

SECONDARY OUTCOMES:
Scale of Prodromal Symptoms - Positive Subscale (SOPS-Pos) | 8 weeks
Global Function: Role scale | 8 weeks
Global Function: Social scale | 8 weeks
Beck Scale for Suicidal Ideation (BSS) | 4 weeks
Calgary Depression Scale for Schizophrenia | 4 weeks
MATRICS Consensus Cognitive Battery (MCCB) | 4 weeks
Relationships Across Domains (RAD) | 4 weeks
Reading the Mind in the Eyes Task (RMET) | 4 weeks
The Awareness of Social Inferences Test (TASIT) | 4 weeks
Emotion Recognition - 40 (ER-40) | 4 weeks
Interpersonal Reactivity Index (IRI) | 4 weeks
Simulator Sickness Questionnaire (SSQ) | 4 weeks
Functional Brain Imaging | 4 weeks
  Change in regional brain activity measured with functional MRI
Structural Brain Imaging | 4 weeks
  Changes in brain structure (e.g., white matter tract integrity) measure with structural MRI

CONTACTS AND LOCATIONS:
Overall Officials: George Foussias, MD PhD FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research